CLINICAL TRIAL: NCT06121388
Title: International Peace Maternity and Child Health Hospital (IPMCH) Affiliated to School of Medicine, Shanghai Jiaotong University, Shanghai, China
Brief Title: Brain MRI Imaging Changes and Associated Factors on Cognition Function in Patients With Premature Ovarian Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Dongmei Lai, Principal Investigator, International Peace Maternity and Child Health Hospital
Other Study IDs: GFY2023007
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Premature Ovarian Failure
Keywords: Premature Ovarian Failure; brain MRI; cognition function
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- health control group: Health control women with similar age, BMI, working environment, education level and regular menstrual cycle in our hospital, and conduct endocrine examination for health examination.
- premature ovarian failure group: Patients are diagnosed with premature ovarian failure.

SUMMARY:
The purpose of this study is to investigate the brain MRI imaging changes and associated factors on cognition function in patients with premature ovarian failure.

DETAILED DESCRIPTION:
Premature Ovarian Failure (POF) refers to a disease characterized by amenorrhea, infertility, low estrogen levels, and high gonadotropin concentration in women before the age of 40. In recent years, the incidence has shown a significant increase. The average age of POF in China is 28.9 years old, involving 2 million women of childbearing age. POF patients have significant emotional disorders and cognitive changes, but it is not known whether the structure and function of the POF patients' brain have changed. It is known that the perimenopause (i.e. estrogen decline) may be the early stage of AD. Therefore, this study aims to use brain imaging technology to explore the changes of brain injury in POF patients with the progression of the disease to achieve early assessment of AD in POF patients. The research work of this project is mainly based on multimodal magnetic resonance imaging technology. For the clinical phenomenon of brain dysfunction in POF patients, it analyzes the changes in brain structure and brain function of POF patients for the first time. Using artificial intelligence brain network analysis method, from the perspective of brain structure and brain function, to determine whether there is microstructural transformation of white matter in POF patients and whether it is related to disease progression and serological indicators. Through the implementation of this project, it provides a basis for brain structure and functional changes for the diagnosis and treatment of POF, and provides a basis for large-scale clinical research to guide clinical formulation of reasonable diagnosis and treatment plans and prognosis evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria for premature ovarian failure:

1. Subjects must meet all the following criteria to be included in the study:
2. Female, between 18 and 40 years old;
3. FSH ≥ 40U/L on two occasions at least four weeks;
4. Sign informed consent. 2. Criteria for the health control group: According to the case control principle, at the same time, the investigators select women with similar age, BMI, working environment, education level and regular menstrual cycle in our hospital, and conduct endocrine examination (FSH <10U/L) for health examination.

Exclusion Criteria:

1. Pregnancy or lactation;
2. Patients with secondary ovarian insufficiency (such as causes of the hypothalamus);
3. Chromosomal karyotype abnormalities (such as Turner syndrome, brittle X syndrome);
4. Any disease that requires immediate blood transfusion;
5. Abuse of alcohol, drugs or drugs (for example, laxatives)
6. Allergies to MRI contrast agents;
7. Accompanied by metal implants, claustrophobia and other magnetic resonance scanning contraindications;
8. Accompanied by serious brain organic diseases, such as epilepsy, stroke, encephalitis, brain trauma, and so on. Nervous system diseases, such as Parkinson's disease, have other cognitive-impacting diseases, or serious somatic diseases such as malignant tumors, acute heart failure, multi-organ failure, and so on.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 premature ovarian failure patients of age 18-40 treated in the International Peace Maternity and Child Health Hospital. 50 women with similar age, BMI, working environment, education level and regular menstrual cycle in our hospital, and conduct endocrine examination for health examination.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain structure | 1 year
  Brain structure will be assessed by MRI.

SECONDARY OUTCOMES:
Follicle-stimulating hormone (FSH) serum level | 1 year
  Follicle-stimulating hormone (FSH) serum level will be tested.
Luteinizing hormone (LH) serum level | 1 year
  Luteinizing hormone (LH) serum level will be tested.
Estradiol (E2) serum level | 1 year
  Estradiol (E2) serum level will be tested.
Testosterone (T) serum level | 1 year
  Testosterone (T) serum level will be tested.
Prolactin (PRL) serum level | 1 year
  Prolactin (PRL) serum level will be tested.
Anti-müllerian hormone (AMH) serum level | 1 year
  Anti-müllerian hormone (AMH) serum level will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Lai, M.D., Principal Investigator — The International Peace Maternity and Child Health Hospital
Locations (1):
- The International Peace Maternity and Child Health Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The public can require the data and protocol from clinicaltrials.gov posted by investigator.
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: Public
URL: http://clinicaltrials.gov

REFERENCES:
- [Background] Brown A, Gervais NJ, Rieck J, Almey A, Gravelsins L, Reuben R, Karkaby L, Rajah MN, Grady C, Einstein G. Women's Brain Health: Midlife Ovarian Removal Affects Associative Memory. Mol Neurobiol. 2023 Nov;60(11):6145-6159. doi: 10.1007/s12035-023-03424-6. Epub 2023 Jul 10. PMID 37423941
- [Background] Zeydan B, Tosakulwong N, Schwarz CG, Senjem ML, Gunter JL, Reid RI, Gazzuola Rocca L, Lesnick TG, Smith CY, Bailey KR, Lowe VJ, Roberts RO, Jack CR Jr, Petersen RC, Miller VM, Mielke MM, Rocca WA, Kantarci K. Association of Bilateral Salpingo-Oophorectomy Before Menopause Onset With Medial Temporal Lobe Neurodegeneration. JAMA Neurol. 2019 Jan 1;76(1):95-100. doi: 10.1001/jamaneurol.2018.3057. PMID 30326011
- [Background] Maki PM, Resnick SM. Effects of estrogen on patterns of brain activity at rest and during cognitive activity: a review of neuroimaging studies. Neuroimage. 2001 Oct;14(4):789-801. doi: 10.1006/nimg.2001.0887. PMID 11554798